CLINICAL TRIAL: NCT06096363
Title: Predictors of High-Flow Nasal Cannula Failure (HFNC) in Patients With Acute Hypoxemic Respiratory Failure (AHRF) Using Echocardiography Parameters
Brief Title: Predictors of HFNC Failure in Patients With AHRF Using Echocardiography Parameters
Acronym: AHRF-ECHO
Status: Completed | Type: Observational
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Wincy Wing-Sze Ng, Associate Consultant, Adult Intensive Care Unit, Queen Mary Hospital, Hong Kong
Other Study IDs: UW 23-086-01
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: Echocardiography; Acute Hypoxemic Respiratory Failure; High Flow Nasal Cannula
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography — Transthoracic Echocardiography to look for evidence of right ventricular (RV) dysfunction and right ventricular-pulmonary arterial (RV-PA) uncoupling.

SUMMARY:
Right ventricular dysfunction (RVD) and right ventricular-pulmonary arterial (RV-PA) uncoupling detected by transthoracic echocardiography (TTE) in acute respiratory distress syndrome (ARDS) are associated with poor survival. Early detection of RVD and RV-PA uncoupling in patients with acute hypoxemic respiratory failure (AHRF) may be indicative of worsening and decompensating pulmonary condition which may require escalation of respiratory support. The use of TTE parameters in predicting high-flow nasal cannula (HFNC) failure has not been previously studied. The objective of this study is to identify predictors of HFNC failure by TTE and to compare its performance with the well-established ROX index.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18; AND
* Acute hypoxemic respiratory failure (AHRF), defined by respiratory rate of greater than 25 breaths per minute and a ratio of the PaO2 to the fraction of inspired oxygen (PaO2 / FiO2) of less than 300, and use of accessory muscles of respiration or paradoxical abdominal motion; AND
* Required ventilatory support with high-flow nasal cannula (HFNC)

Exclusion Criteria:

* Patients suffering from hypercapnic respiratory failure; OR
* AHRF secondary to conditions that are indicated for non-invasive ventilation (NIV) (e.g. acute exacerbation of COPD, cardiogenic pulmonary edema); OR
* Use of NIV or invasive mechanical ventilation (IMV) prior to HFNC initiation; OR
* Patients with imminent need for endotracheal intubation and invasive mechanical ventilation (IMV); OR
* Patients with known or suspected diaphragm paralysis; OR
* Pregnancy; OR
* Patients with abdominal compartment syndrome; OR
* Use of HFNC for more than 12 hours prior to ICU admission; OR
* Patients with suboptimal echocardiographic image quality for data processing; OR

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute hypoxemic respiratory requiring ventilatory support with high flow nasal cannula
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
High-flow nasal cannula (HFNC) therapeutic failure | From the start of recruitment into study (i.e. start of HFNC use), till the date of study endpoint (i.e., step up to non-invasive ventilation, intubation, death on HFNC, or weaned off HFNC, whichever came first), assessed up to 4 weeks.
  Predictive value of transthoracic echocardiography (TTE) in detecting High-flow nasal cannula (HFNC) therapeutic failure in patients with acute hypoxemic respiratory failure (AHRF).

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided